CLINICAL TRIAL: NCT00807755
Title: Phase I Trial of Carboplatin and Etoposide in Combination With Everolimus (RAD001) in Advanced Solid Tumors, With Emphasis on Small Cell Lung Cancer (SCLC)
Brief Title: Everolimus, Carboplatin, and Etoposide in Treating Patients With Small Cell Lung Cancer or Other Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Number of known toxicities observed despite a treatment-naïve population
Sponsor: University of California, Davis (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#214; 200816670 (Other: UC Davis); CRAD001CUS41T (Other: Novartis Pharmaceuticals); UCDCC-214 (Other: University of California, Davis - Cancer Center)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide; etoposide phosphate; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I Dose-Escalation (Experimental): This is a phase I dose escalation study of RAD001 and carboplatin/etoposide. Patients will be accrued in a standard 3 + 3 design based on toxicities experienced during the first cycle. Ten additional chemotherapy naive extensive stage small cell lung cancer (ES-SCLC) patients will be accrued at the Maximum Tolerated Dose (MTD) for further toxicity and response assessment.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: RAD001

INTERVENTIONS:
Drug: Carboplatin — Intravenous (IV) on Day 1 of each 21-day cycle, as per dose escalation schedule (dose levels 1 and 2: dose levels 3 and 4). Number of cycles: 6 maximum.
  Other Names: Paraplatin
Drug: Etoposide — 80mg/m2, Intravenous on Days 1, 2, 3 of a 21-day cycle (all dose levels). Number of cycles: 6 maximum.
  Other Names: Eposin; Etopophos; Vepesid; VP-16
Drug: RAD001 — Orally on Days 1-21 of a 21-day cycle, as per dose escalation schedule (dose level 1: 2.5 mg, dose level 2: 5 mg, dose level 3: 5.0 mg, and dose level 4: 10.0 mg). Number of cycles: unlimited (drug taken from Day 1 until progression of disease or unacceptable toxicity).
  Other Names: Everolimus; Afinitor

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carboplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with everolimus may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus, carboplatin, and etoposide in treating patients with small cell lung cancer or other advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of everolimus combined with carboplatin and etoposide in patients with advanced solid tumors, with emphasis on small cell lung cancer (SCLC).

Secondary

* Determine the maximum-tolerated dose of this regimen in these patients.
* Describe the dose-limiting toxicities and toxicity profile associated with this regimen in these patients.
* Determine, preliminarily, the efficacy of this regimen in an expanded cohort of patients with SCLC.
* Assess the pharmacokinetic parameters of everolimus in this combination.

OUTLINE: This is a dose-escalation study.

Patients receive oral everolimus on days 1-21, carboplatin IV over 15-30 minutes on day 1, and etoposide IV over 30 minutes on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients in the expanded cohort undergo blood collection on days 1, 15, and 22 for pharmacokinetic studies by liquid chromatography-tandem mass spectrometry.

After completion of study therapy, patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumors for which curative standard treatments are not available

  * Ten additional patients with extensive stage small cell lung cancer are accrued to the expanded cohort once a maximum tolerate dose (or a dose for further exploration) is determined

    * Must be chemotherapy naive
* Measurable or evaluable disease

  * Prior irradiated disease sites are considered measurable if there is clear disease progression following radiation therapy
* No uncontrolled brain or leptomeningeal metastases (including those requiring glucocorticoids)

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Life expectancy > 3 months
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.3 mg/dL OR creatinine clearance > 40 mL/min
* Serum bilirubin ≤ 1.5 mg/dL (regardless of liver involvement)
* SGOT ≤ 3 times upper limit of normal (ULN)
* INR ≤ 1.3 (≤ 3 if on anticoagulation)
* Fasting serum cholesterol ≤ 300 mg/dL*
* Fasting triglycerides ≤ 2.5 times ULN*
* No severe and/or uncontrolled medical co-morbidities or other conditions that could affect participation in the study including, but not limited to, the following:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to first study treatment
  * Serious uncontrolled cardiac arrhythmia
  * Severely impaired lung function
  * Active (acute or chronic) or uncontrolled infection
  * Non-malignant medical illness that is uncontrolled or that the control may be jeopardized by the study therapy
  * Liver disease (i.e., cirrhosis, chronic active hepatitis, chronic persistent hepatitis)
* No uncontrolled diabetes mellitus (i.e., fasting serum glucose > 1.5 times ULN)
* No HIV seropositivity
* Not pregnant or nursing
* Fertile patients must use effective contraception

  * No oral, implantable, or injectable contraceptives
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* No active, bleeding diathesis
* No known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
* Must be able to take and retain oral medication
* No peripheral neuropathy > grade 1 as per NCI CTCAE vs. 3 NOTE: *In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid-lowering medication.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* More than 3 weeks since prior and no concurrent investigational drugs
* At least 3 weeks since prior chemotherapy
* At least 2 weeks since prior major surgery or completion of radiotherapy
* No immunization with attenuated live vaccines within the past week or during study therapy
* No prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, or everolimus)
* No chronic treatment with systemic steroids or other immunosuppressive agents
* No concurrent oral anti-vitamin K medication (except low dose coumadin)
* No concurrent medications interfering with everolimus
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of combining RAD001 with carboplatin and etoposide in advanced solid tumors, with emphasis on SCLC. | Up to 1 year from start of treatment

SECONDARY OUTCOMES:
Maximum-tolerated dose as assessed by NCI CTCAE, Version 3.0 | April 2011
Dose-limiting toxicities and toxicity profile as assessed by NCI CTCAE, Version 3.0 | Up to one year.
Preliminary efficacy of this regimen in patients with small cell lung cancer | Up to one year
Pharmacokinetic parameters | Up to one year
Exploratory biomarker analysis | Up to one year

CONTACTS AND LOCATIONS:
Overall Officials: David Gandara, MD, Principal Investigator — University of California School of Medicine - Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States